CLINICAL TRIAL: NCT00240344
Title: REALISTIC: Protocol for an Observational Study in High Risk Patients Switched From Higher Doses of Other Statins to Crestor on the Percentage of Patients Reaching the New EAS LDL-C Target Goal
Brief Title: Study in High Risk Patients Switched From Higher Doses of Other Statins to Crestor on the Percentage of Patients Reaching the New LDL-C Target Goal
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NL401142; REALISTIC
Record Dates: First submitted 2005-10-16; First posted 2005-10-18 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Hypercholesterolemia
Keywords: High risk patients; Crestor; Rosuvastatin; LDL cholesterol; observational
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine the efficacy of Crestor in high risk patients switched from higher doses of other statins in obtaining the new European Atherosclerosis Society (EAS) low-density lipoprotein cholesterol (LDL-C) guidelines.

ELIGIBILITY:
Inclusion Criteria:

* High risk patients
* High doses of other statins
* LDL-C known, starts with Crestor 10 mg
* Permission to use patient data by AstraZeneca (AZ)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care
Sampling Method: Non-Probability Sample
Enrollment: 2650 (Actual)
Dates: Start 2004-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Netherlands Medical Director, MD, Study Director — AstraZeneca
Locations (75):
- Netherlands (75):
  - Research Site, 's-Hertogenbosch
  - Research Site, Alkmaar
  - Research Site, Almelo
  - Research Site, Alphen aan den Rijn
  - Research Site, Amsterdam
  - Research Site, Apeldoorn
  - Research Site, Assen
  - Research Site, Bergen op Zoom
  - Research Site, Beverwijk
  - Research Site, Bilthoven
  - Research Site, Blaricum
  - Research Site, Boxmeer
  - Research Site, Breda
  - Research Site, Brunssum
  - Research Site, Capelle aan den IJssel
  - Research Site, Delft
  - Research Site, Delfzijl
  - Research Site, Den Helder
  - Research Site, Dirksland
  - Research Site, Doetinchem
  - Research Site, Dokkum
  - Research Site, Dordrecht
  - Research Site, Drachten
  - Research Site, Ede Gld
  - Research Site, Eindhoven
  - Research Site, Emmen
  - Research Site, Enschede
  - Research Site, Etten-Leur
  - Research Site, Flushing
  - Research Site, Geldrop
  - Research Site, Gouda
  - Research Site, Groningen
  - Research Site, Haarlem
  - Research Site, Hardenberg
  - Research Site, Heerenveen
  - Research Site, Heerlen
  - Research Site, Helmond
  - Research Site, Hengelo Ov
  - Research Site, Hoofddorp
  - Research Site, Hoogeveen
  - Research Site, Hoorn
  - Research Site, IJmuiden
  - Research Site, Landsmeer
  - Research Site, Leiden
  - Research Site, Lelystad
  - Research Site, Maastricht
  - Research Site, Meppel
  - Research Site, Oosterhout Nb
  - Research Site, Oss
  - Research Site, Purmerend
  - Research Site, Roermond
  - Research Site, Roosendaal
  - Research Site, Rotterdam
  - Research Site, Schiedam
  - Research Site, Sneek
  - Research Site, Spijkenisse
  - Research Site, Stadskanaal
  - Research Site, Terneuzen
  - Research Site, The Hague
  - Research Site, Tiel
  - Research Site, Tilburg
  - Research Site, Utrecht
  - Research Site, Veghel
  - Research Site, Veldhoven
  - Research Site, Venlo
  - Research Site, Vlaardingen
  - Research Site, Waalwijk
  - Research Site, Weert
  - Research Site, Winschoten
  - Research Site, Winterswijk
  - Research Site, Zaandam
  - Research Site, Zevenaar
  - Research Site, Zoetermeer
  - Research Site, Zutphen
  - Research Site, Zwolle